CLINICAL TRIAL: NCT00187915
Title: Pilot Trial for Implementation of a MPA PK Monitoring Strategy
Acronym: MPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEL330; 20030499 (Other: Western Institutional Review Board)
Record Dates: First submitted 2005-09-14; First posted 2005-09-16 (Estimated); Last update posted 2011-10-20 (Estimated); Status verified 2011-10

CONDITIONS: Transplant, Kidney
Keywords: Renal transplant; Cellcept; Therapeutic drug level; Mycophenolate mofetil (MMF); Mycophenolate Acid (MPA); Oral Bioavailability; Immunosuppression
MeSH Terms: interventions — Mycophenolic Acid; Tacrolimus; Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CellCept + Prograf (Other): Standard of Care Regime
  Interventions: Drug: Mycophenolate mofetil + Tacrolimus
- CellCept + Neoral (Other): Standard of Care Regime
  Interventions: Drug: Mycophenolate mofetil + Cyclosporin

INTERVENTIONS:
Drug: Mycophenolate mofetil + Tacrolimus — Target MPA exposure to 30-60 mg/L/h during first month post-transplant
  Other Names: MMF; CellCept; Ro 70-0003; Prograf
  Arms: CellCept + Prograf
Drug: Mycophenolate mofetil + Cyclosporin — Target MPA exposure to 30-60 mg/L/h during first month post-transplant
  Other Names: MMF; CellCept; RO 70-0003; Neoral
  Arms: CellCept + Neoral

SUMMARY:
This study is a prospective interventional trial of de novo renal transplant recipients, aiming to validate a strategy which combines the use of early post transplant MPA AUC sampling, and subsequent MPA trough level monitoring to implement MPA PK monitoring in a clinically applicable fashion.

DETAILED DESCRIPTION:
Mycophenolate mofetil or MMF (CellCept® by Roche) is the mofetil ester of mycophenolic acid (MPA), the active immunosuppressant.

MMF significantly decreases the episodes of acute rejection in kidney transplant patients; but as with any medication without adequate pharmacokinetic drug monitoring, the issue of under or over immunosuppression arises. For this reason, the biggest challenge lies with establishing a feasible mean of MPA pharmacokinetic monitoring. Thus far no study has shown that measuring MPA trough levels alone correlates with rejection, unlike MPA Area Under the concentration time Curve (AUC), due to the large incidence of inter- and intra-patient variability.

This is the first prospective blinded trial set up to analyze the correlation between individualized MPA AUC and trough levels of kidney transplant patients in hopes of establishing a more efficacious way of monitoring MPA. MPA target trough levels that correspond to AUC greater than 30 mg x h/L could then be utilized as maintenance measurements.

ELIGIBILITY:
Inclusion Criteria:

* primary or secondary cadaveric or living donor kidney recipients
* On Cellcept

Exclusion Criteria:

* Multi organ recipients
* Documented non-compliance
* Not on a calcineurin inhibitor
* GFR <25 ml/min by Cockcroft Gault equation
* Serum albumin <2.5 mg/dl
* Pregnant
* Active serious digestive disorder

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2003-07; Primary Completion 2004-11 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Number of subjects with an average AUC between 30-60 ng x hr/mL | 7 months

SECONDARY OUTCOMES:
Rate of acute rejection of transplanted kidney | 7 months
Number of MPA related toxicities | 7 months
Number of dose changes required to obtain MPA AUC target in the first month | 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Herwig-Ulf Meier-Kriesche, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Background] Placebo-controlled study of mycophenolate mofetil combined with cyclosporin and corticosteroids for prevention of acute rejection. European Mycophenolate Mofetil Cooperative Study Group. Lancet. 1995 May 27;345(8961):1321-5. PMID 7752752
- [Background] Sollinger HW. Mycophenolate mofetil for the prevention of acute rejection in primary cadaveric renal allograft recipients. U.S. Renal Transplant Mycophenolate Mofetil Study Group. Transplantation. 1995 Aug 15;60(3):225-32. doi: 10.1097/00007890-199508000-00003. PMID 7645033
- [Background] A blinded, randomized clinical trial of mycophenolate mofetil for the prevention of acute rejection in cadaveric renal transplantation. The Tricontinental Mycophenolate Mofetil Renal Transplantation Study Group. Transplantation. 1996 Apr 15;61(7):1029-37. PMID 8623181
- [Background] Meier-Kriesche HU, Steffen BJ, Hochberg AM, Gordon RD, Liebman MN, Morris JA, Kaplan B. Long-term use of mycophenolate mofetil is associated with a reduction in the incidence and risk of late rejection. Am J Transplant. 2003 Jan;3(1):68-73. doi: 10.1034/j.1600-6143.2003.30112.x. PMID 12492713
- [Background] Meier-Kriesche HU, Steffen BJ, Hochberg AM, Gordon RD, Liebman MN, Morris JA, Kaplan B. Mycophenolate mofetil versus azathioprine therapy is associated with a significant protection against long-term renal allograft function deterioration. Transplantation. 2003 Apr 27;75(8):1341-6. doi: 10.1097/01.TP.0000062833.14843.4B. PMID 12717227
- [Background] Hale MD, Nicholls AJ, Bullingham RE, Hene R, Hoitsma A, Squifflet JP, Weimar W, Vanrenterghem Y, Van de Woude FJ, Verpooten GA. The pharmacokinetic-pharmacodynamic relationship for mycophenolate mofetil in renal transplantation. Clin Pharmacol Ther. 1998 Dec;64(6):672-83. doi: 10.1016/S0009-9236(98)90058-3. PMID 9871432
- [Background] van Gelder T, Hilbrands LB, Vanrenterghem Y, Weimar W, de Fijter JW, Squifflet JP, Hene RJ, Verpooten GA, Navarro MT, Hale MD, Nicholls AJ. A randomized double-blind, multicenter plasma concentration controlled study of the safety and efficacy of oral mycophenolate mofetil for the prevention of acute rejection after kidney transplantation. Transplantation. 1999 Jul 27;68(2):261-6. doi: 10.1097/00007890-199907270-00018. PMID 10440399
- [Background] van Gelder T, Shaw LM. The rationale for and limitations of therapeutic drug monitoring for mycophenolate mofetil in transplantation. Transplantation. 2005 Oct 15;80(2 Suppl):S244-53. doi: 10.1097/01.tp.0000186380.61251.fc. PMID 16251857
- [Background] Shaw LM, Mick R, Nowak I, Korecka M, Brayman KL. Pharmacokinetics of mycophenolic acid in renal transplant patients with delayed graft function. J Clin Pharmacol. 1998 Mar;38(3):268-75. doi: 10.1002/j.1552-4604.1998.tb04424.x. PMID 9549665
- [Background] van Gelder T, Klupp J, Barten MJ, Christians U, Morris RE. Comparison of the effects of tacrolimus and cyclosporine on the pharmacokinetics of mycophenolic acid. Ther Drug Monit. 2001 Apr;23(2):119-28. doi: 10.1097/00007691-200104000-00005. PMID 11294511
- [Background] Srinivas TR, Meier-Kriesche HU, Kaplan B. Pharmacokinetic principles of immunosuppressive drugs. Am J Transplant. 2005 Feb;5(2):207-17. doi: 10.1111/j.1600-6143.2005.00748.x. PMID 15643980
- [Background] Yamani MH, Starling RC, Goormastic M, Van Lente F, Smedira N, McCarthy P, Young JB. The impact of routine mycophenolate mofetil drug monitoring on the treatment of cardiac allograft rejection. Transplantation. 2000 Jun 15;69(11):2326-30. doi: 10.1097/00007890-200006150-00018. PMID 10868634
- [Background] Shaw LM, Pawinski T, Korecka M, Nawrocki A. Monitoring of mycophenolic acid in clinical transplantation. Ther Drug Monit. 2002 Feb;24(1):68-73. doi: 10.1097/00007691-200202000-00012. No abstract available. PMID 11805725
- [Background] Mourad M, Wallemacq P, Konig J, de Frahan EH, Eddour DC, De Meyer M, Malaise J, Squifflet JP. Therapeutic monitoring of mycophenolate mofetil in organ transplant recipients: is it necessary? Clin Pharmacokinet. 2002;41(5):319-27. doi: 10.2165/00003088-200241050-00001. PMID 12036390
- [Background] Cattaneo D, Perico N, Gaspari F, Gotti E, Remuzzi G. Glucocorticoids interfere with mycophenolate mofetil bioavailability in kidney transplantation. Kidney Int. 2002 Sep;62(3):1060-7. doi: 10.1046/j.1523-1755.2002.00531.x. PMID 12164891
- [Background] Shaw LM, Korecka M, Venkataramanan R, Goldberg L, Bloom R, Brayman KL. Mycophenolic acid pharmacodynamics and pharmacokinetics provide a basis for rational monitoring strategies. Am J Transplant. 2003 May;3(5):534-42. doi: 10.1034/j.1600-6143.2003.00079.x. No abstract available. PMID 12752309
- [Background] Cattaneo D, Gaspari F, Ferrari S, Stucchi N, Del Priore L, Perico N, Gotti E, Remuzzi G. Pharmacokinetics help optimizing mycophenolate mofetil dosing in kidney transplant patients. Clin Transplant. 2001 Dec;15(6):402-9. doi: 10.1034/j.1399-0012.2001.150607.x. PMID 11737117
- [Background] Flechner SM, Goldfarb D, Modlin C, Feng J, Krishnamurthi V, Mastroianni B, Savas K, Cook DJ, Novick AC. Kidney transplantation without calcineurin inhibitor drugs: a prospective, randomized trial of sirolimus versus cyclosporine. Transplantation. 2002 Oct 27;74(8):1070-6. doi: 10.1097/00007890-200210270-00002. PMID 12438948